CLINICAL TRIAL: NCT05582421
Title: Effect of Diclofenac Sodium Versus Calcium Hydroxide as Intracanal Medication on the Intensity of Postoperative Pain, Bacterial Load Reduction and MMP-9 Levels in Patients With Necrotic Pulp: A Randomized Clinical Trial
Brief Title: Effect of Diclofenac Sodium Versus Calcium Hydroxide as Intracanal Medication on the Intensity of Postoperative Pain, Bacterial Load Reduction and MMP-9 Levels in Patients With Necrotic Pulp.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohammed awadd, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1141821228
Record Dates: First submitted 2022-10-07; First posted 2022-10-17 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Necrotic Pulp; Apical Periodontitis
Keywords: necrosis
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis; Necrosis | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: Trial Design: Randomized Clinical Trial (Parallel Group) Two Arms Allocation Ratio: 1:1 Framework: Superiority
Who Masked: Participant, Investigator
Masking Description: * In this proposed study, both the participant and assessor will be blinded. This is achieved where the outcome assessor will not be informed of the group in which the participant is enrolled for subjective outcomes. The participants will be blinded to the study hypothesis as to which intervention is expected to be better.
  * The patients who already do not know their treatment group will assess the level of their post-operative pain.
  * The laboratory technician at the microbiological department will not know the treatment group of the patients.
  * The treatment groups will remain anonymous at the end of the study during assessment by the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium hydroxide (Sham Comparator): calcium hydroxide will be placed as intracanal medication between visits.
  Interventions: Drug: Diclofenac Sodium
- diclofenac sodium (Active Comparator): diclofenac sodium will be placed as intracanal medication between visits
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Diclofenac Sodium — intracanal medication

SUMMARY:
the aim of this study is to compare the effect of using Diclofenac Sodium Versus Calcium Hydroxide as Intracanal medication on intensity of postoperative pain, bacterial load reduction after root canal preparation and periapical matrix metalloproteinase 9 level (MMP-9) post-instrumentation and pre-obturation in teeth with necrotic pulp

DETAILED DESCRIPTION:
To compare the effect of diclofenac sodium versus calcium hydroxide as intra canal medication on:

- Primary Outcome Intensity of postoperative pain will be measured using numerical rating scale (NRS) at 6, 12, 24 and 48- hours post-instrumentation and at 6, 12, 24 and 48 hours post-obturation.

Secondary Outcome 1 Bacterial load reduction will be determined by bacterial counting using agar culture technique after root canal preparation (CFU/ml).

Secondary Outcome 2 Periapical MMP-9 level will be determined post-instrumentation and pre-obturation by ELISA.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion criteria:

* Patients who are free from any physical or mental handicapping condition with no underlying systemic disease.
* Age between 18-50 years.
* Males & Females.
* Mandibular single rooted permanent premolar teeth:

  * Diagnosed clinically with pulp necrosis.
  * Absence of spontaneous pain.
  * Positive pain on percussion denoting apical periodontitis.
  * Slight widening in the periodontal membrane space or with periapical radiolucency not exceeding 2*2 mm radiographically.
* Patients' acceptance to participate in the trial.
* Patients who can understand pain scale and can sign the informed consent

Exclusion Criteria:

* Medically compromised patients
* Pregnant women.
* If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively.
* Patients reporting bruxism or clenching.
* Teeth that show association with acute periapical abscess and swelling.
* Greater than grade I mobility or pocket depth greater than 5mm.
* Non-restorable teeth
* Teeth with vital pulp.
* Immature teeth.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
change in Intensity of postoperative pain | 6,12.24.48 hours
  measured using numerical rating scale (NRS) at 6, 12, 24 and 48- hours post-instrumentation and at 6, 12, 24 and 48 hours post-obturation.

SECONDARY OUTCOMES:
Bacterial load reduction | 7 days
  bacterial counting using agar culture technique after root canal preparation (CFU/ml).

OTHER OUTCOMES:
Periapical MMP-9 level | 7 days
  determined post-instrumentation and pre-obturation by ELISA.

IPD SHARING:
Plan to Share IPD: Undecided